CLINICAL TRIAL: NCT02716467
Title: Effect of Intercessory Prayer on the Levels of Psychological Variables, Spiritual and Biological of Patients With Breast Cancer in Radiotherapy Treatment: Clinical Trial
Brief Title: Effect of Intercessory Prayer in Patients With Breast Cancer in Radiotherapy Treatment: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Prado Simão, Student of the Nursing Doctoral, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EERP/USP
Record Dates: First submitted 2016-03-06; First posted 2016-03-23 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: nursing; intercessory prayer; spirituality; clinical trials
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intercessory prayer group (Experimental): Patients in the experimental group receive prayer of intercession during radiotherapy treatment.
  Interventions: Other: intercessory prayer; Radiation: Radiotherapy
- Radiotherapy Treatment (Active Comparator): Patients in the radiotherapy group not receive prayer of intercession during radiotherapy treatment.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Other: intercessory prayer — Intercessory prayer will be offered by a group of six Christian people.
  Arms: intercessory prayer group
Radiation: Radiotherapy — All participants will receive treatment by radiotherapy

SUMMARY:
Living with breast cancer and forms of treatment, among them radiation therapy can cause both side effects such as pain, fatigue and skin changes that affect the well-being, as anxiety, feelings of isolation and changes in routine, which generate existential conflicts and allow the origin of the spiritual anguish phenomenon, which in turn, aggravates the physical and emotional symptoms and the ability to fight the disease. Thus, this study aims to evaluate the effect of intercessory prayer on levels of spiritual distress, religious / spiritual coping, psychological morbidity (anxiety and depression) and amylase levels salivary present in patients with breast cancer radiotherapy.

DETAILED DESCRIPTION:
Reflection on the existence and the meaning of life, common among people with breast cancer radiotherapy generates a suffering that, when directed to the spiritual dimension, results in spiritual distress. In addition, combined with the presence of this phenomenon can flourish during this phase psychological morbidity such as anxiety and depression. In order to face this situation, each person uses cognitive and behavioral strategy according to their beliefs and their meaning of life (religious / spiritual coping). The use of intercessory prayer, where an individual asks a higher being for the benefit of someone seen as receiver, is a strategy that can help people cope with the situation of illness and restore your health. Prayer is one of these activities in the nursing intervention "spiritual support" (5420) proposed by the Nursing Interventions Classification (NIC). a complementary alternative therapy is considered and can be used as an adjuvant in radiotherapy. Therefore, the aim of this study is to verify that the intercession of prayer cause positive effects on levels of spiritual distress, religious coping / spiritual and psychological morbidity (anxiety and depression) present in patients with breast cancer radiotherapy. Thus, a clinical trial will be used randomized controlled and mascaraed. Intervention group will receive the prayer of intercession and control groups (positive and negative) usual care. The data will be analyzed using the Statistical Package for the Social Sciences version 20.0 and will be adopted as the reference value p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with breast cancer in adjuvant and neoadjuvant radiotherapy treatment;
* Both female and male participants are being studiedolder;
* Minimum age of participants is 18 years.

Exclusion Criteria:

* Not being with consciousness, memory and orientation preserved;
* Patients with clinical conditions that affect the continuity in the study or express request not to continue participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07-15 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Spiritual Distress assessed using a scale | an average of 1 year
  spiritual distress

SECONDARY OUTCOMES:
Anxiety and Depression assessed using a scale | an average of 1 year
  anxiety and depression
anxiety assessed per physiological parameter using saliva | an average of 1 year
  anxiety
Short Spiritual Religious Coping assessed using a scale | an average of 1 year
  Short Spiritual Religious Coping

CONTACTS AND LOCATIONS:
Overall Officials: Emília C. Carvalho, PhD, Study Director — Ribeirão Preto College of Nursing
Locations (1):
- Radiotherapy Clinic of the Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No